CLINICAL TRIAL: NCT04227847
Title: A Phase 1 Study of SEA-CD70 in Myeloid Malignancies
Brief Title: A Safety Study of SEA-CD70 in Patients With Myeloid Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SGNS70-101; C5781001 (Other: Alias Study Number); 2023-506945-42-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2020-01-10; First posted 2020-01-14 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Myelodysplastic Syndrome; Acute Myeloid Leukemia
Keywords: Seattle Genetics
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Azacitidine; venetoclax

STUDY DESIGN:
Intervention Model Description: Parts B and C may enroll in parallel after enrollment of Part A is complete. Part D will enroll after Part A is complete. Parts E, F and Part G will enroll in parallel once Part D is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A (Experimental): SEA-CD70 dose escalation cohort in relapsed/refractory (HMA-failure) MDS
  Interventions: Drug: SEA-CD70
- Part B (Experimental): SEA-CD70 expansion cohort in relapsed/refractory (HMA-failure) MDS
  Interventions: Drug: SEA-CD70
- Part C (Experimental): SEA-CD70 expansion cohort in relapsed/refractory AML
  Interventions: Drug: SEA-CD70
- Part D (Experimental): SEA-CD70 + azacitidine dose-finding/dose optimization cohorts in relapsed/refractory MDS or MDS/AML, and previously untreated higher-risk MDS or MDS/AML
  Interventions: Drug: SEA-CD70; Drug: azacitidine
- Part E (Experimental): SEA-CD70 + azacitidine expansion cohort in previously untreated higher-risk MDS or MDS/AML
  Interventions: Drug: SEA-CD70; Drug: azacitidine
- Part F (Experimental): SEA-CD70 + azacitidine expansion cohort in relapsed/refractory MDS or MDS/AML
  Interventions: Drug: SEA-CD70; Drug: azacitidine
- Part G (Experimental): SEA-CD70 + azacitidine +venetoclax dose-finding/dose optimization in previously untreated and unfit for induction therapy AML
  Interventions: Drug: SEA-CD70; Drug: azacitidine; Drug: Venetoclax

INTERVENTIONS:
Drug: SEA-CD70 — Given into the vein (IV; intravenously) on Days 1 and 15 of each treatment cycle
Drug: azacitidine — 75mg/m^2 injected under the skin (SC; subcutaneous) or given into the vein (IV; intravenously) on Days 1 through 7 of each treatment cycle.
  Other Names: VIDAZA
  Arms: Part D; Part E; Part F; Part G
Drug: Venetoclax — 400 mg /day PO, continuously; administered with ramping
  Other Names: Venclexta
  Arms: Part G

SUMMARY:
This trial will look at a drug called SEA-CD70 with and without azacitidine, to find out if it is safe for participants with myelodysplastic syndrome (MDS) and acute myeloid leukemia (AML). It will study SEA-CD70 to find out what its side effects are and if it works for AML and MDS. A side effect is anything the drug does besides treating cancer.

This study will have seven groups or "parts."

* Part A will find out how much SEA-CD70 should be given to participants
* Part B will use the dose found in Part A to find out how safe SEA-CD70 is and if it works to treat participants with MDS.
* Part C will use the dose found in Part A to find out how safe SEA-CD70 is and if it works to treat participants with AML.
* Part D will find out how much SEA-CD70 with azacitidine should be given to participants
* Part E will use the dose found in Part D to find out how safe SEA-CD70 with azacitidine is and if it works to treat participants with MDS or MDS/AML that has not been treated.
* Part F will use the dose found in Part D to find out how safe SEA-CD70 with azacitidine is and if it works to treat participants with MDS or MDS/AML.
* Part G will find out how much SEA-CD70 with azacitidine and with venetoclax should be given to participants with AML. Also, to evaluate safety and tolerability of PF-08046040 in combination with azacitidine and venetoclax in participants with previously untreated AML who are unfit for standard induction chemotherapy.

DETAILED DESCRIPTION:
This is a phase 1, open-label, multicenter, dose-finding, and dose expansion study designed to evaluate the safety, tolerability, pharmacokinetics (PK), and antitumor activity of SEA-CD70 monotherapy and SEA-CD70 in combination with azacitidine in adults with myeloid malignancies. The study will be conducted in up to 6 parts.

* Part A is a dose-escalation cohort designed to identify the MTD or recommended expansion dose of SEA-CD70 monotherapy in participants with relapsed/refractory (hypomethylating agent [HMA]-failure) MDS.
* Part B is an expansion cohort designed to evaluate the safety and tolerability of SEA-CD70 monotherapy in participants with relapsed/refractory (HMA-failure) MDS.
* Part C is an expansion cohort designed to evaluate the safety and tolerability of SEA-CD70 monotherapy in participants with relapsed/refractory AML.
* Part D contains dose-finding/dose optimization cohorts designed to evaluate the safety/tolerability and identify the recommended expansion dose of SEA-CD70 in combination with azacitidine in participants with 1) relapsed/refractory (HMA-failure) MDS or MDS/AML, and 2) previously untreated higher-risk per IPSS-M (Moderate High, High or Very High) MDS or MDS/AML.
* Part E is an expansion cohort designed to evaluate the safety and tolerability of SEA-CD70 in combination with azacitidine in participants with previously untreated higher-risk per IPSS-M (Moderate High, High, or Very High) MDS or MDS/AML.
* Part F is an expansion cohort designed to evaluate the safety and tolerability of SEA-CD70 in combination with azacitidine in participants with relapsed/refractory (HMA-failure) MDS or MDS/AML.
* Part G will find out how much SEA-CD70 with azacitidine and with venetoclax should be given to participants with previously untreated AML who are unfit for standard of care induction chemotherapy

ELIGIBILITY:
Part A Inclusion Criteria

* Participants with cytologically/histologically confirmed MDS (2016 World Health Organization (WHO) classification) with

  * Measurable disease per WHO MDS with excess blasts criteria
  * MDS that is relapsed or refractory and must not have other therapeutic options
  * Treatment failure after prior hypomethylating agent (HMA) therapy for MDS
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1

Part B Inclusion Criteria

* Participants with cytologically/histologically confirmed MDS (WHO classification) with:

  * Measurable disease per WHO MDS with excess blasts (MDS-EB) criteria
  * MDS that is relapsed or refractory and must not have other therapeutic options
  * Treatment failure after prior HMA therapy for MDS
* ECOG Performance Status of 0-2

Part C Inclusion Criteria

* Participants with relapsed or refractory AML (ICC 2022) (except for acute promyelocytic leukemia [APL]):

  * Who have received either 2 or 3 previous regimens
  * Who have received 1 previous regimen to treat active disease and have at least one of the following:

    * Age > 60 and ≤75 years.
    * Primary resistant AML or secondary AML
    * First CR duration <6 months
    * Adverse-risk per European Leukemia Network genetic risk stratification
* Age 18-75 years
* ECOG performance status of 0-2

Parts D and F Inclusion Criteria

* Participants with diagnosis of MDS or MDS/AML (ICC 2022 criteria)
* Disease which has relapsed, failed to respond after minimum of 6 cycles, or progressed following an HMA in the immediately preceding line of therapy.
* Eligible for continued therapy with azacitidine
* ECOG Performance Status 0-2

Parts D and E Inclusion Criteria

* Participants with diagnosis of MDS or MDS/AML (ICC 2022 criteria), previously untreated.
* Participants with higher-risk per IPSS-M MDS and MDS/AML
* ECOG Performance Status 0-2

Part G Inclusion Criteria

* Participants with diagnosis of AML (ICC 2022 criteria), previously untreated and ineligible for standard induction chemotherapy.
* Age ≥18 years.
* ECOG Performance Status of 0-2.

Exclusion Criteria (All Parts)

* Previous exposure to CD70-targeted agents
* Prior allogeneic hematopoietic stem cell transplant, for any condition
* Central nervous system leukemia
* History of clinically significant sickle cell anemia, autoimmune hemolytic anemia, or idiopathic thrombocytopenic purpura
* Parts D, F and G only: Prior oral HMA or oral HMA-combinations
* Part G: conditions that preclude enteral route of administration; concomitant use of strong/moderate CYP3A inducers; history of myeloproliferative neoplasm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2020-08-07 (Actual); Primary Completion 2027-07-04 (Estimated); Study Completion 2028-07-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Through 30-37 days following last dose of SEA-CD70; up to approximately 2 years
  Any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Number of participants with laboratory abnormalities | Through 30-37 days following last dose of SEA-CD70; up to approximately 2 years
  To be summarized using descriptive statistics.
Number of participants with a dose-limiting toxicity (DLT) at each dose level (Parts A and D only) | Though end of DLT evaluation period; up to approximately 4 weeks
  To be summarized using descriptive statistics.

SECONDARY OUTCOMES:
AUC - Area under the plasma concentration-time curve | Through 30-37 days following last dose of SEA-CD70; up to approximately 2 years
  To be summarized using descriptive statistics.
Tmax - Time to maximum concentration attained | Through 30-37 days following last dose of SEA-CD70; up to approximately 2 years
  To be summarized using descriptive statistics.
Cmax - Maximum observed plasma concentration | Through 30-37 days following last dose of SEA-CD70; up to approximately 2 years
  To be summarized using descriptive statistics.
Ctrough - Minimum plasma concentration per dosing interval | Through 30-37 days following last dose of SEA-CD70; up to approximately 2 years
  To be summarized using descriptive statistics.
T1/2 - Terminal elimination half-life | Through 30-37 days following last dose of SEA-CD70; up to approximately 2 years
  To be summarized using descriptive statistics.
Incidence of antidrug antibodies (ADA) | Through 30-37 days following last dose of SEA-CD70; up to approximately 2 years
  To be summarized using descriptive statistics.
Complete remission (CR) Rate and complete remission equivalent (CReq) rate | Up to approximately 4 years
  Proportion of participants with AML, MDS/AML or MDS who achieve CR or CReq
Complete remission with incomplete blood count recovery (CRi) rate | Up to approximately 4 years
  Proportion of participants with AML who achieve CRi
Complete remission with limited count recovery (CRL) rate for participants with MDS or MDS/AML | Up to approximately 4 years
  Proportion of participants with MDS or MDS/AML who achieve CRL
Complete remission with partial hematologic recovery (CRh) rate | Up to approximately 4 years
  Proportion of participants with AML, MDS/AML, or MDS who achieve CRh
Hematologic response (HI) rate | Up to approximately 4 years
  Proportion of participants with MDS or MDS/AML with HI
Overall response rate (ORR) | Up to approximately 4 years
  For AML, the proportion of participants who achieve a best response of CR, CRi, CRh, or partial response (PR). For MDS, the proportion of participants who achieve a best response of CR, CReq, CRL, CRh, PR, or HI
Duration of remission (DOR) | Up to approximately 4 years
  For AML, the time from first CR/CRi/CRh/PR response to the first documentation of disease progression, start of new anticancer therapy, or death due to any cause. For MDS, the time from first CR (or Req)/CRL/CRh/PR to the first documentation of disease progression, start of new anticancer therapy, or death due to any cause
Overall survival (OS) | Up to approximately 4 years
  Time from start of study treatment to the date of death due to any cause
Event-free survival (EFS) | Up to approximately 4 years
  Time from first dose to the first documentation of progression, failure to achieve remission within 6 months of study entry, disease relapse, or death due to any cause, whichever comes first.
Progression-free survival (PFS) | Up to approximately 4 years
  Time from first dose to the first documentation of progression, disease relapse, or death from any cause, whichever comes first
MRD-negative ORR | Up to approximately 4 years
  Proportion of participants with AML or MDS who achieve MRD-negative ORR
Time to response (TTR) | Up to approximately 4 years
  Time from start of study treatment to the first documentation of objective response
Rate of conversion to transfusion independence (TI) | Up to approximately 4 years
  Proportion of participants who convert from transfusion dependence at baseline to TI post-baseline
Rate of TI maintenance | Up to approximately 4 years
  Proportion of participants who were TI at baseline and maintain TI post-baseline

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (53):
- United States (48):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Dept. of Medicine, UAB ONeal Comprehensive Cancer Center, Birmingham, Alabama
  - City of Hope (City of Hope National Medical Center, City of Hope Medical Center), Duarte, California
  - IP Address: City of Hope Investigational Drug Services(IDS), Duarte, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Hematology-Oncology Clinic, Los Angeles, California
  - Colorado Blood Cancer Institute, Lab, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian/St. Luke's Medical Center, Denver, Colorado
  - The University of Kansas Cancer Center ,Investigational Drug Services, Fairway, Kansas
  - The University of Kansas Clinical Research Center, Fairway, Kansas
  - The University of Kansas Hospital, Kansas City, Kansas
  - University of Kansas Hospital Cambridge North Tower A, Kansas City, Kansas
  - University of Kansas Medical center Medical office building, Kansas City, Kansas
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - The University of Kansas Cancer Center - Overland Park, Overland Park, Kansas
  - The University of Kansas Cancer Center - Indian Creek Campus, Overland Park, Kansas
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Norton Hospitals, Inc, Louisville, Kentucky
  - Norton Cancer Institute, St. Matthews Campus, Attn. Becky Champion, PharmD, Louisville, Kentucky
  - Norton Cancer Institute, St. Matthews Campus, Louisville, Kentucky
  - Norton Women & Children's Hospital, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber/Mass General Brigham Cancer Care, Inc, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer Institute Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - The University of Kansas Cancer Center - Medical Oncology Clinic, Kansas City, Missouri
  - The University of Kansas Cancer Center - Radiation Oncology Clinic, Kansas City, Missouri
  - The University of Kansas Cancer Center -North, Kansas City, Missouri
  - The University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Columbia University Irving Medical Center, New York, New York
  - CUIMC Research Pharmacy, New York, New York
  - The New York and Presbyterian Hospital, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center/James Cancer Hospital, Columbus, Ohio
  - Hollings Cancer Center, Charleston, South Carolina
  - Medical University of South Carolina- Ashley River Tower, Charleston, South Carolina
  - Medical University of South Carolina- Investigational Drug Services, Charleston, South Carolina
  - Medical University of South Carolina- University Hospital, Charleston, South Carolina
  - Baylor Research Institute, Dallas, Texas
  - Baylor University Medical Center, Investigational Drug Services, Department of Pharmacy, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
- Japan (3):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - Yamagata University Hospital, Yamagata
- Netherlands (2):
  - Pharmacy - UMC Utrecht t.a.v. Apotheek KGO, Utrecht
  - University Medical Center (UMC) Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Dewulf J, Flieswasser T, Delahaye T, Vangestel C, Miranda A, de Haard H, Jacobs J, Smits E, Van den Wyngaert T, Elvas F. Site-specific 68Ga-labeled nanobody for PET imaging of CD70 expression in preclinical tumor models. EJNMMI Radiopharm Chem. 2023 Apr 24;8(1):8. doi: 10.1186/s41181-023-00194-3. PMID 37093350
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=SGNS70-101